CLINICAL TRIAL: NCT01571024
Title: A Phase I Study of BKM120 With mFOLFOX6 in Patients With Advanced Solid Tumors With Expansion Cohort in Metastatic Pancreatic Cancers.
Brief Title: BKM120 + mFOLFOX6 in Advanced Solid Tumors With Expansion Cohort Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1036
Record Dates: First submitted 2012-01-03; First posted 2012-04-04 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Advanced Solid Tumors; Metastatic Colorectal Cancer; Metastatic Pancreatic Cancer
Keywords: FOLFOX6; BKM120; Advanced Solid Tumors; Metastatic; Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — NVP-BKM120; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 + mFOLFOX6 (Experimental): BKM120 + mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer.
  Interventions: Drug: BKM120; Drug: mFOLFOX6

INTERVENTIONS:
Drug: BKM120 — BKM120 40 mg, orally, once daily.
  Other Names: buparlisib
Drug: mFOLFOX6 — mFOLFOX6 treatment will be as follows: Oxaliplatin: 85 mg/m2 IV, Leucovorin: 400 mg/m2 IV, 5FU bolus: 400 mg/m2 IV and 5FU infusion: 2400 mg/m2 IV.
  Other Names: Folinic acid (leucovorin); Fluorouracil (5-FU); Oxaliplatin (Eloxatin)

SUMMARY:
The purpose of this study is to establish the safety and tolerability of BKM120 when combined with mFOLFOX6 and to define the maximum tolerated dose of BKM120 in this combination in advanced solid tumors including metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This single arm, multicenter, open-label Phase I clinical trial has been designed to establish the safety and tolerability of dose escalating BKM120 when combined with mFOLFOX6 and to define the MTD of BKM120 in this combination. Secondary objective will be to estimate the response rate, Progression Free Survival rate, and Overall Survival rate, after treatment with the Maximum Tolerated Dose of BKM120 in combination with mFOLFOX6 in patients with advanced solid tumors and metastatic pancreatic cancer. Eligible patients will be treated with BKM120 orally (PO), once per day (QD) in combination with mFOLFOX6 administered intravenously (IV) every 2 weeks on Days 1 and 15 of each cycle using a standard 3+3 dose escalation scheme. Each cycle will be repeated every 4 weeks (28 days). FOLFOX6 treatment will be as follows: Oxaliplatin: 85 mg/m2 IV, Leucovorin: 400 mg/m2 IV, 5FU bolus: 400 mg/m2 IV and 5FU infusion: 2400 mg/m2 IV.

In the absence of treatment delays due to adverse events (AEs), treatment may continue until: disease progression, intercurrent illness that prevents further administration of treatment, unacceptable AE(s), patient decides to withdraw from the study, or general or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Age ≥18 years (no upper age limit)
2. Histologically confirmed advanced solid tumor that is refractory to standard therapy or for which there is no accepted standard therapy. In the initial determination of the MTD, any solid tumor type is acceptable. For the expansion cohort 15 patients with untreated metastatic pancreatic cancer.
3. Measurable or nonmeasurable (but evaluable) disease as determined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) for determination of the MTD. Measurable disease is required for the expansion cohort.
4. Patients must have normal organ and marrow function as defined below: Absolute neutrophil count ≥1,500/μL, Platelets ≥100,000/μL, Hemoglobin > 9g/dL (transfusion allowed), Total bilirubin within normal range, or ≤1.5 X upper limit of normal (ULN) if liver metastases are present; or total bilirubin ≤3 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome. AST(SGOT)/ALT(SGPT) within normal limits (WNL), except for patients with tumor involvement of the liver who must have AST and ALT ≤3 X ULN Serum creatinine ≤1.5 X ULN OR 24-hour creatinine clearance ≥60 mL/min Amylase and lipase levels WNL Fasting plasma glucose ≤120 mg/dL (7.8 mmol/L), INR ≤2.
5. Total calcium (corrected for serum albumin) WNL (bisphosphonate use for malignant hypercalcemia control is not allowed).
6. Brain metastases permitted if: CNS-directed treatment has been given; Off CNS-directed therapy >3 months; AND CNS disease has been clinically and radiographically stable for at least 8 weeks and patient not receiving corticosteroid therapy
7. Life expectancy ≥12 weeks
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
9. No limit to prior number of cytotoxic chemotherapies provided time since the last dose of prior therapy (in advance of Day 1 of study treatment): Cytotoxic chemotherapy ≥ the duration of the most recent cycle of the previous regimen (with a minimum of 4 weeks for all, except minimum of 6 weeks for nitrosourea, mitomycin-C) Biologic therapy (e.g. antibodies) ≥4 weeks ≥5 X half-life of a small molecule therapeutic (e.g. tyrosine kinase inhibitor [TKI])
10. Ability to understand and willingness to sign a written informed consent document
11. Women of childbearing potential (WOCBP) and all men must be willing and able to use appropriate contraception (double barrier method); WOCBP must have negative pregnancy test within 72 hours before Day 1 of treatment.
12. Patient must have recovered from all reversible toxicities related to their previous treatment except for alopecia and grade 1 neuropathy

Exclusion Criteria:

1. Patients with history of prior treatment with a PI3K inhibitor
2. Patients may not be receiving any other investigational agents currently, or within time limits specified above prior to study Day 1.
3. Patients with known coagulopathies, and those who require therapeutic anti-coagulation with coumarin-derivative anticoagulants
4. Patients on strong or moderate CYP3A4 inhibitor(s) or CYP3A4 inducer(s) unable or unwilling to discontinue during the study period (see Appendix B for list). Please note that co-treatment with weak inhibitors of CYP3A4 is allowed.
5. Patients who received live vaccines or who have close contact with people who have received live vaccines within 7 days of day 1 of BKM120 (see Appendix B).
6. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pomelos, or exotic citrus fruits.
7. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤2 weeks prior to starting study drug. Erythropoietin or darbepoietin therapy, if initiated ≥2 weeks prior to enrollment, may be continued.
8. Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to table 12B for a list of prohibited QT-prolonging drugs with risk of Torsades de Pointes.
9. Patients on chronic steroids (or other immunosuppressive agents) unable or unwilling to discontinue. Note: Topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airway diseases), eye drops, or local injections (e.g., intra-articular) are allowed. Also, short course of corticosteroid for use as an anti-emetic prior to/during chemotherapy, or if needed to manage pneumonitis is allowed.
10. Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
11. Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire: Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicide/homicidal ideation (immediate risk of doing harm to others)) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug. ≥CTCAE Grade 3 anxiety, Meets the cut-off score of ≥ 10 on the 9-item Patient Health Questionnaire (PHQ-9) or a cut-off score of ≥15 on the 7-item, Generalized Anxiety Disorder (GAD-7) mood scale, or who selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study unless overruled by the psychiatric assessment.
12. Patients with diarrhea CTCAE v4 grade ≥2
13. Patient having active cardiac disease including any of the following: Left ventricular ejection fraction (LVEF) <50% as determined by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO), QTc >480 msec on screening ECG (using the QTcF formula), Angina pectoris that requires the use of anti-anginal medication, Ventricular arrhythmias except for benign premature ventricular contractions, Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication, Conduction abnormality requiring a pacemaker Valvular disease with documented compromise of cardiac function, Symptomatic pericarditis.
14. Patient having a history of cardiac dysfunction including any of the following: Myocardial infraction within the last 6 months documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function, History of documented congestive heart failure (CHF) by New York Heart Association (NYHA) functional classification III-IV, Documented cardiomyopathy.
15. Known diagnosis of human immunodeficiency virus (HIV) infection
16. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection. Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, carbon monoxide diffusing capacity (DLco), and O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates.
17. Impaired GI function or GI disease that may significantly impair absorption of BKM120 (e.g., irritable bowel disease [IBD] malabsorption syndrome, small bowel resection, uncontrolled vomiting, or diarrhea).
18. Patients who have received wide field radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
19. Patients who have undergone major surgery ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
20. History of allergic reaction attributed to compounds of similar chemical or biologic composition to BKM120, 5FU, leucovorin, or oxaliplatin.
21. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator
22. Grade ≥2 neuropathy at baseline
23. History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix.
24. Pregnant or lactating women or adults of reproductive potential not employing an effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 3 years
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications, and occurs within the first cycle of therapy (4 weeks)of BKM120 when administered with mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer.
Maximum Tolerated Dose (MTD) | 3 years
  The MTD is defined as a dose with a Dose Limiting Toxicity rate of 20% for BKM120 when administered with mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer.

SECONDARY OUTCOMES:
Number of subjects experiencing adverse events | 3 years
  Using CTCAE criteria, we will identify acute and chronic toxicities of BKM120 in combination with mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer
Progression Free Survival (PFS) | 4 years
  The length of time subject's disease does not get worse from time of start of treatment with BKM120 in combination with mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer.
Overall Survival(OS) | 7 years
  Length of survival after treatment with the MTD of BKM120 in combination with mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer.
Biomarkers of Clinical Benefit | 3 years
  To examine potential correlations between blood and tissue biomarkers and clinical benefit of BKM120 when administered with mFOLFOX6 in patients with advanced solid tumors including metastatic pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Autumn McRee, MD, Principal Investigator — University of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center; Chapel Hill, NC
Locations (1):
- University of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Website — http://unclineberger.org